CLINICAL TRIAL: NCT04545255
Title: The Use of Low Intensity Shock Wave Therapy for the Treatment of Provoked Vestibulodynia Disorder (PVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, i_gruenwald, Professor, Director of the Neuro- urology unit, Rambam healthcare campus, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0098-18-rmc
Record Dates: First submitted 2020-08-20; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Provoked Vestibulodynia

STUDY DESIGN:
Intervention Model Description: A double-blinded, randomized, sham-controlled, prospective study
Who Masked: Participant, Investigator
Masking Description: Shockwave probes were either active or sham (by blocking energy transfer from probe)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active (Active Comparator): A shockwave device with a probe that conveys shockwave energy
  Interventions: Device: Shockwave treatment
- sham (Sham Comparator): A shockwave device with specially designed probe which has the shockwave energy blocked
  Interventions: Device: Shockwave treatment

INTERVENTIONS:
Device: Shockwave treatment — ED 1000 shockwave generator

SUMMARY:
Provoked vestibulodynia (PVD) is an exhausting pain syndrome that immensely affects quality of sexual life, and consequently negatively affects quality of life. Low intensity shock wave therapy produces physical forces that lead to pain relief.

Aim: To evaluate the feasibility, safety and efficacy of low-intensity shockwave therapy in patients with provoked vestibulodynia.

Methods: A double-blinded, randomized, sham-controlled, prospective study of 32 women. The treatment protocol included a series of treatments, performed twice a week for 6 weeks. Each treatment consisted of 500 pulses of low intensity shockwaves (0.09 mJ/〖mm〗^2 ) using the "Medispec ED-1000®" shock wave generator or sham.

DETAILED DESCRIPTION:
The study was a single center, double-blinded, randomized, sham-controlled, prospective study. Study eligibility criteria were treatment at the Neuro-urology Unit in Rambam Medical Center, during January 2018 - January 2020 and a diagnosis of PVD. PVD diagnosis was based on description of the pain and on a positive cotton swab test15.

Women were randomized at a 2:1 ratio to treatment or sham groups. The treatment protocol included a series of treatments, performed twice a week for 6 weeks, for a total of 12 sessions. Each treatment consisted of 500 pulses of low intensity shockwaves (0.09 millijoul/〖mm〗^2 ) using the "Medispec ED-1000®" shock wave generator. The sham protocol included the same treatment protocol without shock wave generator activation. The patients were evaluated three times throughout the trial by an investigator blinded to the group allocation: before the first treatment, and one and three months after the twelfth treatment. Pain was assessed by both subjective and objective measures. The primary outcome measure was a change in dyspareunia, as assessed by scores on the 10-point visual analogue scale (VAS) (range 0-10 ).

Secondary outcome measures for evaluating pain were increases in pain threshold and tolerance, assessed by a quantitative validated algometer test16, 17, the Wong-Baker pain FACES scale (range 0-10)18, the Female Sexual Function Index (FSFI) (range 2-38)19 and the Patients' Global Impression of Change scale (PGIC) (first component range 0-7; 0=no change, 7=a great deal better; second component range 0-10; 0=much better and 10=much worse)20. The PGIC assessed the self-reported impression of a general change due to the intervention.

The algometer applied was a very basic and simple device that was assembled and used at our unit after validating its safety, accuracy, and adequacy in evaluating introitus pain vs control (doctorate dissertation). For assessing the pain threshold with the algometer, radial pressure (mmHg) was applied by progressively inflating a cylindrical balloon inserted in the introitus. The participant was required to report the first painful sensation, and this pressure, defined as the threshold pressure, was registered. The measurement was performed sequentially 4 times and the average of the measured pressures was considered the first pain threshold). Finally, for pain tolerance measurement, the participant was again asked to report when she had reached her pain limit (1-10 on the verbal scale ) upon continuous pressure

ELIGIBILITY:
Inclusion Criteria:

* Above age 18 years
* Diagnosis of provoked vestibulodynia by a gynecologist at least 3 month prior to study date
* Positive cotton swab test
* Pain during intercourse/ tampon insertion, gynecologic examination
* Cognitively and physically adapted for undergoing treatment

Exclusion Criteria:

* Pregnancy or lactating
* History of pelvic or external genitalia irradiation during the past year
* Any chronic neurological disorder causing local pain
* Any pelvic inflammatory process
* Any psychiatric disorders
* Investigators impression of patient being eligible for the study (non compliance etc..)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 1 year
  The primary outcome was a change in dyspareunia, as assessed by scores on the 10-point Visual Analogue Scale where 1 is the minimum score meaning painless and 10 is the maximum score meaning excruciating pain

SECONDARY OUTCOMES:
Algometer testing | 1 year
  measures threshold of pain in mmHg, where any threshold below 100 mmHg is considered pathological
Wong-Baker pain FACES scale | 1 year
  from a scale of 1 to five showing sad face for score 1 and very happy face for score 5
Female Sexual Function Index (FSFI) | 1 year
  A validated questionnaire assessing female sexual dysfunction, any score above 22.5 is pathological
Patients' Global Impression of Change scale. | 1 year
  one question with a scale from -3 to+3 where 0 is not better nor worse, -3 is much worse and +3 is much better

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Healthcare Campus, Haifa, Northern District, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Landry T, Bergeron S, Dupuis MJ, Desrochers G. The treatment of provoked vestibulodynia: a critical review. Clin J Pain. 2008 Feb;24(2):155-71. doi: 10.1097/AJP.0b013e31815aac4d. PMID 18209522
- [Result] Sutton KS, Pukall CF, Chamberlain S. Pain, psychosocial, sexual, and psychophysical characteristics of women with primary vs. secondary provoked vestibulodynia. J Sex Med. 2009 Jan;6(1):205-14. doi: 10.1111/j.1743-6109.2008.01038.x. PMID 19170850